CLINICAL TRIAL: NCT03126773
Title: A Prospective Multicenter Non-interventional Cohort Study on Patients'Satisfaction With Angeliq® Micro in Real Clinical Practice Conducted in Russia
Brief Title: A Prospective Multicenter Study on Patients'Satisfaction With Angeliq® Micro in Real Clinical Practice Conducted in Russia
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 19022
Record Dates: First submitted 2017-04-20; First posted 2017-04-24 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Menopause
Keywords: non-interventional; cohort; Angeliq Micro; menopause; Russia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BAY86-4891: The patients will be treated according to the routine practice. All the patients meeting the criteria of inclusion and exclusion to whom administration of Angeliq Micro is indicated are fit for participation in this non-interventional study.
  Interventions: Drug: BAY86-4891

INTERVENTIONS:
Drug: BAY86-4891 — Drospirenone 0.25 mg + estradiol hemihydrate 0.5 mg (Angeliq Micro, G03FA17).Dosage form is one tablet a day.

SUMMARY:
To evaluate the patients' satisfaction with Angeliq Micro in real clinical practice after 13 cycles of treatment.

DETAILED DESCRIPTION:
This non-interventional study is planned with the aim of obtaining information about the results of the product use in real clinical practice by means of the evaluation of the patients' satisfaction.

The study will be multicenter, non-interventional, prospective, cohort study in patients for whom their physicians have taken a decision about Angeliq Micro treatment, irrespectively of the fact of this study inclusion.

The absence of a control group (patients who receive another menopausal hormonal therapy medication, or do not receive menopausal hormonal therapy at all) is based on high risk of bias (heterogeneity of exposure in case of comparison of low-dosed and ultralow-doses menopausal hormonal therapy regiments, or in case of comparison with a group of patients for whom the menopausal hormonal therapy is not indicated).

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged 50 to 65 years with vasomotor symptoms of menopause (moderate or severe in intensity), who has been prescribed or will be prescribed the menopausal hormonal therapy with Angeliq Micro.
* Patients, who are already receiving continuous combined menopausal hormonal therapy (except Angeliq) for 3-5 years willing to continue MHT, and who will change their therapy for Angeliq Micro.
* Patients who never ever received menopausal hormonal therapy, if at least 3 years have passed after the last menstruation, with the STRAW+10 stage +1c and younger than 60 years at the moment of inclusion.
* Signed informed consent form (written consent for the study participation).

Exclusion Criteria:

* Unwillingness or inability to give the informed consent for the study participation.
* Contraindications for menopausal hormonal therapy (according to the Angeliq Micro SmPC).
* Current use or history of use during 1 month before of dietary supplements containing St John's wort, as they can affect tolerability and safety of hormonal therapy.
* Current participation in any other clinical study

Ages: 50 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Female patients aged 50 to 65 years with vasomotor symptoms of menopause
Sampling Method: Probability Sample
Enrollment: 1570 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-06-18 (Actual)

PRIMARY OUTCOMES:
Patient's satisfaction with the menopausal symptoms treatment after 13 cycles of treatment | Up to 14 months
  Menopause Symptoms Treatment Satisfaction Questionnaire (MS-TSQ) will be considered continuous variable and reported using denoted descriptive statistics. Apart from this, patient's satisfaction will be dichotomised and analysed / reported as "satisfied / not satisfied".

SECONDARY OUTCOMES:
Patient's satisfaction with the menopausal symptoms treatment after 3-4 cycles of treatment | Up to 4 months
  Menopause Symptoms Treatment Satisfaction Questionnaire (MS-TSQ) will be considered continuous variable and reported using denoted descriptive statistics. Apart from this, patient's satisfaction will be dichotomised and analysed / reported as "satisfied / not satisfied".
Changes in menopause symptoms | Up to 14 months
  Menopause Rating Scale (MRS) questionnaire, will be derived from MRS questionnaire at baseline and at subsequent visits (as difference V2-V1 and V3-V1) and reported using denoted descriptive statistics.
Changes in the quality of life | Up to 14 months
  Menopause Rating Scale (MRS) questionnaire, will be derived from MRS questionnaire at baseline and at subsequent visits (as difference V2-V1 and V3-V1) and reported using denoted descriptive statistics.
Approaches to menopausal hormonal therapy prescription | Up to 24 months
  Approaches to menopausal hormonal therapy prescription will be considered discrete variable and reported using denoted descriptive statistics.
Reasons of choice of a low-dosed or ultralow-dosed menopausal hormonal therapy | Up to 24 months
  Reasons of choice of a low-dosed or ultralow-dosed menopausal hormonal therapy will be considered discrete variable and reported using denoted descriptive statistics.
Patients' compliance | Up to 24 months
  Patients' compliance will be considered continuous variable and reported using denoted descriptive statistics.
Number of early discontinuation during the first year of therapy | Up to 12 months
  Early discontinuation during the first year of therapy of Angeliq Micro will be considered binary.
Timing of discontinuation of Angeliq® Micro | Up to 24 months
  Timing of discontinuation of Angeliq Micro will be considered right-censored time-to-event
Reasons of discontinuation of Angeliq Micro | Up to 24 months
  Reasons of discontinuation of Angeliq Micro will be considered multinomial type.
Tolerability of Angeliq Micro in real clinical practice by using MS-TSQ questionnaire | Up to 24 months
  Tolerability of Angeliq Micro will be assessed as question 7 of MS-TSQ questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Many locations, Multiple Locations, Russia

REFERENCES:
- See also: Click here to find results for studies related to Bayer products — http://clinicaltrials.bayer.com/